CLINICAL TRIAL: NCT01386515
Title: The Role of Family Functioning in Promoting Adaptation in Siblings of Individuals With Duchenne Muscular Dystrophy (DMD)
Status: Terminated | Type: Observational
Sponsor: National Human Genome Research Institute (NHGRI) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 999911177; 11-HG-N177
Record Dates: First submitted 2011-06-30; First posted 2011-07-01 (Estimated); Last update posted 2019-12-12 (Actual); Status verified 2016-01-07

CONDITIONS: Genetic Disease; Communication
Keywords: Adaptation; Duchenne Muscular Dystrophy; Communication about Duchenne Muscular Dystrophy; Sibling
MeSH Terms: conditions — Genetic Diseases, Inborn; Communication; Muscular Dystrophy, Duchenne

STUDY DESIGN:
Time Perspective: Other

SUMMARY:
Background:

We want to learn more about the relationship between the way families function and how children adapt to having a sibling with Duchenne muscular dystrophy (DMD). What we learn will help us design better interventions for families.

Objective:

* To learn more about how families with an individual with DMD function.
* To learn how siblings adapt in families with an individual with DMD.

Eligibility:

* One parent and one child, age 13-18, from a family where another child has DMD.
* The parent and the child must be able to read and write English.

Design:

* One parent from each family will complete a survey about how family members communicate and relate with each other. The parent will also answer questions about the behavior of the child without DMD. This survey will take you about 40 minutes to complete.
* One child from each family, either a boy or a girl, will also complete a survey. This survey asks about how he/she views him/herself. It also asks about how he/she interacts with peers and family members and how he/she behaves. The survey also asks how satisfied he/she is with how his/her family functions. This survey takes about 30 minutes to finish.

DETAILED DESCRIPTION:
This study proposes to explore the role of family functioning in promoting adaptation in unaffected siblings of children with Duchenne muscular dystrophy (DMD). Although evidence suggests that family functioning may be a predictor of adaptation in caregivers of children with chronic illnesses, little research has been conducted on the relationships between aspects of family functioning and the adaptation of unaffected siblings. Evidence in the literature suggests that aspects of family functioning may play a key role in adaptation. Moreover, the role of DMD-specific communication in facilitating sibling adaptation has not yet been explored in the literature and further insight may be derived from exploring this relationship. The goals of this study are to better understand the relationship of family functioning with the adaptation of unaffected siblings, as well as to explore the timing, extent (depth and content), and the characteristics of initiation of discussion of parent-sibling communication around DMD. Currently, some evidence exists to direct the creation of interventions that reinforce a family-centered approach to facilitate adaptation of family members to living with a child with a chronic health condition. Nevertheless, more insight is needed to understand how family processes affect individual adaptation, especially that of the unaffected sibling, in order to maximize the effectiveness of future interventions with this population.

ELIGIBILITY:
* INCLUSION CRITERIA:

Parents/Caregivers:

* Parent or caregiver of child with DMD and child without DMD
* Lives with child that does not have DMD
* 18 or older
* Reads/Writes English

Siblings:

* Sibling of child with DMD
* Lives in same household as individual with DMD
* 13-18 years of age
* Reads/Writes English

Min Age: 13 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 33 (Actual)
Dates: Start 2011-06-07; Study Completion 2016-01-07

PRIMARY OUTCOMES:
adaptation, behavior problems, self-concept, pro-social behavior

CONTACTS AND LOCATIONS:
Overall Officials: Barbara B Biesecker, Principal Investigator — National Human Genome Research Institute (NHGRI)
Locations (1):
- National Human Genome Research Institute (NHGRI), 9000 Rockville Pike, Bethesda, Maryland, United States

REFERENCES:
- [Background] Branstetter JE, Domian EW, Williams PD, Graff JC, Piamjariyakul U. Communication themes in families of children with chronic conditions. Issues Compr Pediatr Nurs. 2008 Oct-Dec;31(4):171-84. doi: 10.1080/01460860802475184. PMID 19021037
- [Background] Bushby K, Finkel R, Birnkrant DJ, Case LE, Clemens PR, Cripe L, Kaul A, Kinnett K, McDonald C, Pandya S, Poysky J, Shapiro F, Tomezsko J, Constantin C; DMD Care Considerations Working Group. Diagnosis and management of Duchenne muscular dystrophy, part 2: implementation of multidisciplinary care. Lancet Neurol. 2010 Feb;9(2):177-89. doi: 10.1016/S1474-4422(09)70272-8. Epub 2009 Nov 27. PMID 19945914
- [Background] Chen JY, Clark MJ. Family function in families of children with Duchenne muscular dystrophy. Fam Community Health. 2007 Oct-Dec;30(4):296-304. doi: 10.1097/01.FCH.0000290542.10458.f8. PMID 17873636